CLINICAL TRIAL: NCT06837311
Title: Medical Benefit of Digital Monitoring Using apTeleCare for Secondary Prevention in Patients With a Recent Transient Ischemic Attack or Stroke
Brief Title: Post-Stroke Secondary Prevention With Digital Monitoring
Acronym: PSDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2023/74
Record Dates: First submitted 2025-02-04; First posted 2025-02-20 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: Ecological Momentary Assessment (EMA); Biological: Biological assessment; Behavioral: Psychological examination and Substance Use symptomatology; Other: Treatment as usual (TAU); Diagnostic Test: Expired carbon monoxide (CO)
- Treatment as usual (Other)
  Interventions: Biological: Biological assessment; Behavioral: Psychological examination and Substance Use symptomatology; Other: Treatment as usual (TAU); Diagnostic Test: Expired carbon monoxide (CO)

INTERVENTIONS:
Device: Ecological Momentary Assessment (EMA) — Daily ecological momentary assessment (EMA), in addition to treatment as usual (TAU) using apTeleCare eHealth device. Daily surveys includes questions reflecting all Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 symptom criteria for Depression, Generalized Anxiety Disorder, Post-Traumatic Symptom Disorder, evaluations of substance use (including dietary items at risk) as well as of two symptoms predictive of relapse (craving and loss of control), medication compliance and physical activity
  Arms: Intervention
Biological: Biological assessment — Routine Biological assessment and of substance use
Behavioral: Psychological examination and Substance Use symptomatology — Substance use symptomatology ; Neuropsychiatric symptomatology ; Functional outcomes ; Neurologic and Cardiovascular outcomes
Other: Treatment as usual (TAU) — Treatment as usual (TAU)
Diagnostic Test: Expired carbon monoxide (CO) — Expired carbon monoxide (CO) measurement

SUMMARY:
Stroke is the second leading cause of death and a major cause of disability worldwide. In 2019, Disability-Adjusted Life-Years (DALYs) related to stroke was estimated to have reached 143 million. Modifiable stroke risk-factors, which include poor lifestyle habits (tobacco, alcohol and illicit drug abuse, dietary patterns at risk, low physical activity), account for 90 % of the risk of stroke. Stroke complications and the risk of stroke recurrence is highly dependent on the control of these risk factors. Thus, the secondary prevention of stroke requires profound lifestyle modifications including substance use cessation and diet changes. National guidelines for stroke clinical practice advocate an immediate cessation of consumption of all substances but without recommendations on specific therapeutic regimens. Moreover, none address the management of poor coping with stress or mood problems though they are major population attributable risk factors of stroke and constitute major barriers of behavior changes achievement. Yet, post-stroke emotional impairments are frequent, post-stroke depression and anxiety being the most frequent (prevalence is 30% and 25%, respectively). Importantly, independently from stroke, emotional impairments or disorders and Substance Related and Addiction Disorders (SRADs) are frequent comorbid conditions (dual disorders) with debilitating consequences and the interplay between the two conditions makes rehabilitation more complex. This suggests that taking into account stroke patients' mental health status might improve not only the management of post-stroke emotional impairments but also the control of stroke vascular risk factors.

Regarding secondary prevention programs focusing on behavioral changes among Cardiovascular and Cerebrovascular Disease (CVD) patients, the literature is sparse and studies on smoking cessation are the most widely documented. Despite the risk of smoking after a myocardial infarct or a stroke/Transient Ischemic Attack (TIA), less than half of patients quit smoking after the event or achieve long-term abstinence.

To increase treatment adherence and efficacy, besides systematically screening lifestyle habits and evaluating the patients' mental health and motivation to change in clinical routine, experts in the domain emphasize the need to:

* start delivering treatment as early as possible, ideally during hospitalization;
* tailor the intensity of the treatment (combination of pharmacological medications +/- behavioral intervention; frequency of the follow-up/contacts) according to the risk profile of each patient, particularly depending on the level of dependence and the presence of comorbid emotional difficulties/psychiatric disorders.

After hospital discharge, in standard care, the follow-up visit is scheduled 4 to 6 months post-stroke. Knowing that the vast majority of smoking relapses occur in the weeks following stroke, it appears that this period is of high risk for missing the goal of stroke secondary prevention. Therefore, new approaches are urgently needed that would allow for the day-to-day examination of clinical change in the immediate days and weeks following discharge from the stroke acute-care unit to optimize the patient's recovery and quality of life.

The potential pivotal role of eHealth development has been advocated by the World Health Organization, which considers e-Health as a cost-effective and secure use of information and communication technologies (ICT). Used in the context of stroke secondary prevention, eHealth technologies should give each patient the opportunity to describe his/her own experiences and symptoms and the contexts of daily life in which they occur that may constitute negative factors for post-stroke recovery. Post-stroke management would thus be optimized through a person-centered, intense and multidisciplinary care program.

Investigators believe apTeleCare would allow for such a day-to-day examination of clinical change in the immediate days and weeks following discharge from the stroke acute-care unit. It offers the possibility not only to closely monitor patients' experiences and symptoms and the contexts of daily life in which they occur, but also to inform the clinical team in real-time via specific alerts that depend on the type and level of difficulties the patients encounter for adopting the expected changes in their lifestyle

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 18 years of age and younger than 80 years;
* Recent (≤ 15 days) clinically symptomatic ischemic or hemorrhagic stroke documented through brain imaging (CT or MRI) or a Transient Ischemic Attack with an Predictive Risk Score (ABCD2) ≥ 4;
* Returning to the neurovascular unit for the standard care post-stroke follow-up visits;
* National Institute Health Stroke Scale (NIHSS) < 15;
* modified Rankin scale ≤ 4;
* No severe cognitive impairment as defined by the neurologist;
* Current smokers (smoking at least 1 cigarette per day during the month before admission)
* Able to use a smartphone
* Living in an area with internet coverage
* Written informed consent by the patient;
* Coverage by the French National Health Insurance

Exclusion Criteria:

* Subarachnoid hemorrhage; Dementia syndrome or other central neurologic disorder;
* Severe aphasia (NIHSS item 9 ≥ 2)
* Severe visual impairment interfering with the completion of evaluations;
* Severely impaired physical and/or mental health that, according to the neurologist, may affect the participant's capacity to participate in the study;
* Individuals already undergoing treatment for tobacco cessation and/or SRADs at admission in the stroke unit;
* Pregnancy or breastfeeding;
* Inability to read French;
* Individuals under legal protection or unable to express personally their consent
* Participation in another protocol modifying the patient's follow-up status.
* Person deprived of liberty
* Person in emergency situation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2028-03-25 (Estimated)

PRIMARY OUTCOMES:
Expired carbon monoxide (CO) rate | 6 months
  Prevalence tobacco abstinence (Expired CO ≤ 8 ppm) 6 months after acute ward discharge.

SECONDARY OUTCOMES:
Level of risk and prevalence of Substance-related and addictive disorders (SRADs) | Day 0
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). It consists of 8 questions covering tobacco, alcohol, cannabis, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, opiates, and 'other drugs. Twenty-eight domains/scores are derived from these questions
Level of risk and prevalence of Substance-related and addictive disorders (SRADs) | 3 Months
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). It consists of 8 questions covering tobacco, alcohol, cannabis, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, opiates, and 'other drugs. Twenty-eight domains/scores are derived from these questions
Level of risk and prevalence of Substance-related and addictive disorders (SRADs) | 6 Months
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). It consists of 8 questions covering tobacco, alcohol, cannabis, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, opiates, and 'other drugs. Twenty-eight domains/scores are derived from these questions
Level of risk and prevalence of Substance-related and addictive disorders (SRADs) | 12 Months
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). It consists of 8 questions covering tobacco, alcohol, cannabis, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, opiates, and 'other drugs. Twenty-eight domains/scores are derived from these questions
Fagerström Test for Nicotine Dependence (FTND) score | Day 0
  Nicotine dependence using the Fagerström Test for Nicotine Dependence (FTND) which includes 10 items. Scores can range from 0 to 10. The recommended cut-off scores to index the categories of nicotine dependence severity are as follows: below 2 = no dependence, 3 to 4 = mild severity, 5 to 6 = moderate severity, 7 to 10 = extreme severity.
Fagerström Test for Nicotine Dependence (FTND) score | 3 months
  Nicotine dependence using the Fagerström Test for Nicotine Dependence (FTND) which includes 10 items. Scores can range from 0 to 10. The recommended cut-off scores to index the categories of nicotine dependence severity are as follows: below 2 = no dependence, 3 to 4 = mild severity, 5 to 6 = moderate severity, 7 to 10 = extreme severity.
Fagerström Test for Nicotine Dependence (FTND) score | 6 months
  Nicotine dependence using the Fagerström Test for Nicotine Dependence (FTND) which includes 10 items. Scores can range from 0 to 10. The recommended cut-off scores to index the categories of nicotine dependence severity are as follows: below 2 = no dependence, 3 to 4 = mild severity, 5 to 6 = moderate severity, 7 to 10 = extreme severity.
Fagerström Test for Nicotine Dependence (FTND) score | 12 months
  Nicotine dependence using the Fagerström Test for Nicotine Dependence (FTND) which includes 10 items. Scores can range from 0 to 10. The recommended cut-off scores to index the categories of nicotine dependence severity are as follows: below 2 = no dependence, 3 to 4 = mild severity, 5 to 6 = moderate severity, 7 to 10 = extreme severity.
modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) score | Day 0
  Includes one question to assess each of the 11 DSM 5 diagnostic criteria for SRADs transposed to food items as well as two questions to assess clinically significant distress and impairment. Food Addiction is mild if there are 2 or 3 symptoms and clinically significant impairment/distress, moderate if there are 4 or 5 symptoms and significant impairment/distress, and severe if there are 6 or more symptoms and significant impairment/distress.
modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) score | 3 Months
  Includes one question to assess each of the 11 DSM 5 diagnostic criteria for SRADs transposed to food items as well as two questions to assess clinically significant distress and impairment. Food Addiction is mild if there are 2 or 3 symptoms and clinically significant impairment/distress, moderate if there are 4 or 5 symptoms and significant impairment/distress, and severe if there are 6 or more symptoms and significant impairment/distress.
modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) score | 6 Months
  Includes one question to assess each of the 11 DSM 5 diagnostic criteria for SRADs transposed to food items as well as two questions to assess clinically significant distress and impairment. Food Addiction is mild if there are 2 or 3 symptoms and clinically significant impairment/distress, moderate if there are 4 or 5 symptoms and significant impairment/distress, and severe if there are 6 or more symptoms and significant impairment/distress.
modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) score | 12 Months
  Includes one question to assess each of the 11 DSM 5 diagnostic criteria for SRADs transposed to food items as well as two questions to assess clinically significant distress and impairment. Food Addiction is mild if there are 2 or 3 symptoms and clinically significant impairment/distress, moderate if there are 4 or 5 symptoms and significant impairment/distress, and severe if there are 6 or more symptoms and significant impairment/distress.
Alcohol Use Disorder Identification Test (AUDIT) Score | Day 0
  Alcohol dependence test. 10 items. Scores can range from 0 to 40. The recommended cut-off scores to index the categories of alcohol dependence severity are as follows: from 6 to 12 for women and 7 to 12 for men = moderate severity, and above 12 = extreme severity for both sexes.
Alcohol Use Disorder Identification Test (AUDIT) Score | 3 months
  Alcohol dependence test. 10 items. Scores can range from 0 to 40. The recommended cut-off scores to index the categories of alcohol dependence severity are as follows: from 6 to 12 for women and 7 to 12 for men = moderate severity, and above 12 = extreme severity for both sexes.
Alcohol Use Disorder Identification Test (AUDIT) Score | 6 months
  Alcohol dependence test. 10 items. Scores can range from 0 to 40. The recommended cut-off scores to index the categories of alcohol dependence severity are as follows: from 6 to 12 for women and 7 to 12 for men = moderate severity, and above 12 = extreme severity for both sexes.
Alcohol Use Disorder Identification Test (AUDIT) Score | 12 months
  Alcohol dependence test. 10 items. Scores can range from 0 to 40. The recommended cut-off scores to index the categories of alcohol dependence severity are as follows: from 6 to 12 for women and 7 to 12 for men = moderate severity, and above 12 = extreme severity for both sexes.
Cannabis Abuse Screening Test (CAST) score | Day 0
  6 items. Scores can range from 0 to 6. The recommended cut-off scores to index the categories of cannabis dependence severity are as follows: below 2 = low risk of dependence, a score of 2 = moderate risk of dependence, and 3 or more = high risk of dependence.
Cannabis Abuse Screening Test (CAST) score | 3 Months
  6 items. Scores can range from 0 to 6. The recommended cut-off scores to index the categories of cannabis dependence severity are as follows: below 2 = low risk of dependence, a score of 2 = moderate risk of dependence, and 3 or more = high risk of dependence.
Cannabis Abuse Screening Test (CAST) score | 6 Months
  6 items. Scores can range from 0 to 6. The recommended cut-off scores to index the categories of cannabis dependence severity are as follows: below 2 = low risk of dependence, a score of 2 = moderate risk of dependence, and 3 or more = high risk of dependence.
Cannabis Abuse Screening Test (CAST) score | 12 Months
  6 items. Scores can range from 0 to 6. The recommended cut-off scores to index the categories of cannabis dependence severity are as follows: below 2 = low risk of dependence, a score of 2 = moderate risk of dependence, and 3 or more = high risk of dependence.
Readiness Ruler or Substance Use Motivation Ruler score | Day 0
  Asks the respondent to rank his/her motivation to end his/her substance use on a Visual Analog Scale from 1 (Absolutely no motivation to quit) to 10 (No doubt about the decision to be sober) and to list some motivations. The participant will be instructed to provide at least one motivation or more if relevant.
Readiness Ruler or Substance Use Motivation Ruler score | 3 months
  Asks the respondent to rank his/her motivation to end his/her substance use on a Visual Analog Scale from 1 (Absolutely no motivation to quit) to 10 (No doubt about the decision to be sober) and to list some motivations. The participant will be instructed to provide at least one motivation or more if relevant.
Readiness Ruler or Substance Use Motivation Ruler score | 6 months
  Asks the respondent to rank his/her motivation to end his/her substance use on a Visual Analog Scale from 1 (Absolutely no motivation to quit) to 10 (No doubt about the decision to be sober) and to list some motivations. The participant will be instructed to provide at least one motivation or more if relevant.
Readiness Ruler or Substance Use Motivation Ruler score | 12 months
  Asks the respondent to rank his/her motivation to end his/her substance use on a Visual Analog Scale from 1 (Absolutely no motivation to quit) to 10 (No doubt about the decision to be sober) and to list some motivations. The participant will be instructed to provide at least one motivation or more if relevant.
Hospital Anxiety and Depression scale (HAD) score | Day 0
  assesses the perceived level of depressive (7 items) and anxiety (7 items). For each subscale, a score of 7 or more is considered indexing depression and anxiety caseness.
Hospital Anxiety and Depression scale (HAD) score | 3 Months
  assesses the perceived level of depressive (7 items) and anxiety (7 items). For each subscale, a score of 7 or more is considered indexing depression and anxiety caseness.
Hospital Anxiety and Depression scale (HAD) score | 6 Months
  assesses the perceived level of depressive (7 items) and anxiety (7 items). For each subscale, a score of 7 or more is considered indexing depression and anxiety caseness.
Hospital Anxiety and Depression scale (HAD) score | 12 Months
  assesses the perceived level of depressive (7 items) and anxiety (7 items). For each subscale, a score of 7 or more is considered indexing depression and anxiety caseness.
Multidimensional Assessment of Thymic States scale (MAThYS) Score | Day 0
  visual analog scale of 20 items relating to individual states as perceived by the patient for the preceding week. Items can be grouped into five quantitative dimensions ranging each from inhibition to excitation: 1. emotional reactivity, 2. thought processes, 3. psychomotor function, 4. Motivation, and 5. sensory perception
Multidimensional Assessment of Thymic States scale (MAThYS) Score | 3 Months
  visual analog scale of 20 items relating to individual states as perceived by the patient for the preceding week. Items can be grouped into five quantitative dimensions ranging each from inhibition to excitation: 1. emotional reactivity, 2. thought processes, 3. psychomotor function, 4. Motivation, and 5. sensory perception
Multidimensional Assessment of Thymic States scale (MAThYS) Score | 6 Months
  visual analog scale of 20 items relating to individual states as perceived by the patient for the preceding week. Items can be grouped into five quantitative dimensions ranging each from inhibition to excitation: 1. emotional reactivity, 2. thought processes, 3. psychomotor function, 4. Motivation, and 5. sensory perception
Multidimensional Assessment of Thymic States scale (MAThYS) Score | 12 Months
  visual analog scale of 20 items relating to individual states as perceived by the patient for the preceding week. Items can be grouped into five quantitative dimensions ranging each from inhibition to excitation: 1. emotional reactivity, 2. thought processes, 3. psychomotor function, 4. Motivation, and 5. sensory perception
Checklist for Cognitive and Emotional Consequences following stroke (CLCE-24) score | Day 0
  standardized instrument that includes 13 cognitive items, 9 emotional items, and 2 additional open-ended, non-specified items concerning potential additional difficulties not evaluated by the other items. The scoring of each item ranges from 0 (not present) to 3 (present and affecting daily life).
Checklist for Cognitive and Emotional Consequences following stroke (CLCE-24) score | 3 Months
  standardized instrument that includes 13 cognitive items, 9 emotional items, and 2 additional open-ended, non-specified items concerning potential additional difficulties not evaluated by the other items. The scoring of each item ranges from 0 (not present) to 3 (present and affecting daily life).
Checklist for Cognitive and Emotional Consequences following stroke (CLCE-24) score | 6 Months
  standardized instrument that includes 13 cognitive items, 9 emotional items, and 2 additional open-ended, non-specified items concerning potential additional difficulties not evaluated by the other items. The scoring of each item ranges from 0 (not present) to 3 (present and affecting daily life).
Checklist for Cognitive and Emotional Consequences following stroke (CLCE-24) score | 12 Months
  standardized instrument that includes 13 cognitive items, 9 emotional items, and 2 additional open-ended, non-specified items concerning potential additional difficulties not evaluated by the other items. The scoring of each item ranges from 0 (not present) to 3 (present and affecting daily life).

CONTACTS AND LOCATIONS:
Overall Officials: Igor SIBON, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided